CLINICAL TRIAL: NCT04747678
Title: Tolerability and Adverse Effects of Using Multiple Doses of Ivermectin in Egypt During Covid 19 Pandemic
Brief Title: Adverse Effects of Ivermectin Used in Egypt During COVID-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, ahmed mohamed esmat fahim mansour, Principal Investigator, Menoufia University
Other Study IDs: ahmed19782020
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Covid19; Ivermectin Poisoning; Drug Toxicity; Drug Side Effect
MeSH Terms: conditions — COVID-19; Drug-Related Side Effects and Adverse Reactions | interventions — Ivermectin

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days

INTERVENTIONS:
Drug: Ivermectin — retrograde study of common and rare adverse effects of multiple doses of ivermectin used during the coivd 19 pandemic in egypt

SUMMARY:
retrograde study of common and rare adverse effects of multiple doses of ivermectin used during the coivd 19 pandemic in egypt

DETAILED DESCRIPTION:
ivermectin was used in Egypt during the pandemic of covid-19 and it was registered in the MOH protocol that has been published in November 2020 the study will document the adverse effects of many patients used ivermectin as aprophylaxis and as a treatment with multiple dose regimens

ELIGIBILITY:
Inclusion Criteria:

* all people used ivermectin as a treatment or as a prophylactic in covid 19 pandemic in egypt with explained dose

Exclusion Criteria:

-

Ages: 16 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all healthy and diseased people who used ivermectin the last three months either as a treatment or as a prophylaxis with mention of the doses used and the adverse effects experienced during and after the usage
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-03 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
all adverse effects will be collected from people used Ivermectin in between September 2020 to December 2020 | the data will be collected from February 2021 to march 2021
  all data will be collected from retrospective manner as a retrospective study

SECONDARY OUTCOMES:
all data will be arranged according to time and dose manner | February to match 2021
  data for each dose will be identified together

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mansour, Shibīn al Kawm, Menoufia, Egypt